CLINICAL TRIAL: NCT03350997
Title: Effects of Exercise and Energy Balance on 24-hour Blood Glucose Control
Acronym: CGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, Associate Professor, Movement Science, School of Kinesiology, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00120520
Record Dates: First submitted 2017-11-13; First posted 2017-11-22 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Metabolic Disease; Adipose Tissue
Keywords: Exercise
MeSH Terms: conditions — Metabolic Diseases; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial 1 (Experimental): Subjects will have two CGM devices placed on either side of the abdomen, near the belly button. Trial 1 Exercise - subjects will use a mouthpiece and nose clip (which will allow all of their expired air to pass through the metabolic cart for analysis of oxygen consumption and carbon dioxide production) for ~5 min at the beginning, middle and toward the end of exercise to verify they are exercising at 65% of VO2peak. This will allow us to accurately measure energy expenditure (kcal) during exercise. One hour after the exercise session, participants will eat a standardized dinner which includes the energy expended from their exercise session (+ 350 kcal).
  Interventions: Behavioral: Trial 1 Exercise
- Trial 2 (Experimental): Subjects will have one CGM device placed on one side of the abdomen. Trial 2 Exercise - subjects will exercise at 65% of VO2peak. One hour after the exercise session, participants will eat a standardized dinner which will NOT include the energy expended from their exercise session (- 350 kcal).
  Interventions: Behavioral: Trial 2 Exercise

INTERVENTIONS:
Behavioral: Trial 2 Exercise — During the exercise session, subjects will exercise at 65% of VO2peak. One hour after the exercise session, participants will eat a standardized dinner which will NOT include the energy expended from their exercise session (- 350 kcal).
  Arms: Trial 2
Behavioral: Trial 1 Exercise — During the exercise session, subjects will use a mouthpiece and nose clip (which will allow all of their expired air to pass through the metabolic cart for analysis of oxygen consumption and carbon dioxide production) for ~5 min at the beginning, middle and toward the end of exercise to verify they are exercising at 65% of VO2peak. This will allow us to accurately measure energy expenditure (kcal) during exercise. One hour after the exercise session, participants will eat a standardized dinner which includes the energy expended from their exercise session (+ 350 kcal).
  Arms: Trial 1

SUMMARY:
The study team will assess "free-living" 24h glucose control using continuous glucose monitors (CGM) over an 88h period on two separate occasions. Importantly, standardized meals will be provided and will be consumed at specific times each day of the CGM measurement period. These meals will be identical on day 1 and day 3 of measurement. Each subject will complete two CGM periods, which will be identical except for the calorie and macronutrient content of the post-exercise dinner. In addition, during trial 1, two CGM's will be worn, while only 1 CGM will be worn on trial 2.

DETAILED DESCRIPTION:
Subjects will be instructed to exercise exactly 2 days before each experimental trial period, and then abstain from exercise other than the exercise session on Day 2 of the trial period until after the trial period is complete.

Subjects will arrive to the Substrate Metabolism Laboratory at approximately 4pm on Day 0 of each trial. For trial 1, two CGM devices will be placed on either side of the abdomen, near the belly button. For trial 2, only one CGM device will be placed on one side of the abdomen.

On Day 1 of both trials, participants will go about their normal daily activities (other than planned exercise) while eating provided meals at designated time points. This day will serve as the non-exercise control day.

On Day 2, subjects will return to the laboratory to exercise on the bike for ~1h at a moderate exercise intensity (approximately 65% of their measured VO2peak) to expend 350 kilocalories. During trial 1 only, subjects will use the mouthpiece and nose clip (which will allow all of their expired air to pass through the metabolic cart for analysis of oxygen consumption and carbon dioxide production) for ~5 min at the beginning, middle and toward the end of exercise to verify they are exercising at 65% of VO2peak. This will also allow the study team to accurately measure energy expenditure (kcal) during exercise. On trial 2, subjects will perform the exact same exercise protocol, but the mouthpiece and nose clip will not be required. One hour after the exercise session, participants will eat their standardized dinner. Importantly, the caloric content of this meal will differ between the two trials (+/- 350kcal), and this will be the only difference between the two study trial periods.

On Day 3, participants will go about their normal daily activities (other than planned exercise) while eating the provided meals at designated time points. This day will serve as the post-exercise day.

On Day 4, participants will return to the laboratory at approximately 8am for removal of the CGM device(s).

ELIGIBILITY:
Inclusion criteria

* Age: 18-40
* Body Mass Index: 20-30 kg/m2

Exclusion criteria

* Pregnant or lactating
* Evidence/history of cardiovascular or metabolic disease
* Medications known to affect glucose metabolism

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Average Post-prandial glucose values | 1 week
  Average Post-prandial glucose values (1 hour, 2 hour, and 3 hours) will be measured
area under curve Post-prandial glucose values (1 hour, 2 hour, and 3 hours) | 1 week
  1 hour, 2 hour, and 3 hours time-point for Post-prandial glucose values will be measured

SECONDARY OUTCOMES:
24 hour glycemic response | 1 day
  Average 24 hour glycemic response will be measured
Area under curve - 24 hour glycemic response | 1 day
  24 hour glycemic response area under curve will be measured
CGM Sensor Variability when measured simultaneously | 1 week
  coefficient variation of blood glucose between the 2 CGM devices placed during trial 1

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Horowitz, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States